CLINICAL TRIAL: NCT01176981
Title: Assessing the Safety, Feasibility, Cost Effectiveness and Patient Satisfaction of Outpatient Administration of High Dose Methotrexate (HD MTX) in Patients With Osteosarcoma
Brief Title: Outpatient Administration of High Dose Methotrexate (HD MTX) in Patients With Osteosarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Abha Gupta, Staff Physician, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000018144
Record Dates: First submitted 2010-08-03; First posted 2010-08-06 (Estimated); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Osteosarcoma
Keywords: pediatrics; Osteosarcoma; Methotrexate; Outpatient
MeSH Terms: conditions — Osteosarcoma | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HDMTX (Experimental): This is a single arm study. All subjects enrolled in the study will be in this arm.
  Interventions: Drug: High Dose Methotrexate

INTERVENTIONS:
Drug: High Dose Methotrexate — Methotrexate will be given by IV at a dose of 12 gram/m2/dose.
  The patient will receive 4-6 hours of hydration with alkalinization, and then HD MTX will be infused over 4 hours. Following this, the patient will be discharged home to receive continuous intravenous hydration through a portable pump. The patient will return to hospital daily for a comprehensive clinical assessment, IV hydration and antiemetics, MTX level and creatinine monitoring until MTX is cleared (3-4 days).

SUMMARY:
The primary purpose of this study is to determine the safety and feasibility of delivering HDMTX in an outpatient setting.

DETAILED DESCRIPTION:
High Dose Methotrexate (HDMTX) is an integral part of osteosarcoma therapy whose main toxicities include myelosuppression, mucositis, nephrotoxicity, and hepatitis. In order to deliver HDMTX therapy safely, patients require urinary alkalinization, hydration, monitoring of renal function, therapeutic drug monitoring, and leucovorin rescue. Due to the required supportive care needs, HDMTX has historically been given as an inpatient. In some centers however, HDMTX is being given safely as an outpatient in order to reduce health care costs, improve patient quality of life and to deliver timely therapy with limited inpatient chemotherapy beds available.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 years of age;
* Localized or metastatic osteosarcoma;
* Adequate renal function (GFR > 70 ml/1.73m2) prior to each cycle;
* No grade III/IV renal toxicity, mucositis or vomiting with most recent prior inpatient MTX cycle;
* Parent and/or patient must be able to provide written consent, and complete Patient Flow Sheets in English.

Exclusion Criteria:

* Patients, in the opinion of the primary healthcare team, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal.
* Pregnant females
* Breastfeeding females

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abha Gupta, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29965827/

RESULTS

PARTICIPANT FLOW:
Groups:
- HDMTX: This is a single arm study. All subjects enrolled in the study will be in this arm.
  High Dose Methotrexate: Methotrexate will be given by IV at a dose of 12 gram/m2/dose.
  The patient will receive 4-6 hours of hydration with alkalinization, and then HD MTX will be infused over 4 hours. Following this, the patient will be discharged home to receive continuous intravenous hydration through a portable pump. The patient will return to hospital daily for a comprehensive clinical assessment, IV hydration and antiemetics, MTX level and creatinine monitoring until MTX is cleared (3-4 days).
Period: Overall Study
Arm/Group | HDMTX
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | HDMTX
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 13.5 [10 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: The Number of Outpatient High Dose Methotrexate Courses Which Result in an Inpatient Hospital Admission.
Description: Patients will be evaluated prior to and daily during each outpatient HDMTX course, and if one or more of a list of hospitalization criteria are met, the patient will be admitted to hospital to complete that course.
Time Frame: 9 months
Measure: Number; unit: courses of MTX
Units Other Than Participants: courses of MTX
Groups:
- HD MTX: all patients received outpatient HD MTX
Arm/Group | HD MTX
Number analyzed (Participants) | 6
Number analyzed (courses of MTX) | 72
courses of MTX | 0

ADVERSE EVENTS:
Arm/Group | HDMTX
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No